CLINICAL TRIAL: NCT04640376
Title: Comparison of the Analgesic Effect of a New Paracetamol Formulation (Paracetamol UNIFLASH) for Buccal Use and Two Different Doses of an Oral Paracetamol Form Controlled Versus Placebo in Patients Suffering From Moderate Pain Due to a Tooth Extraction.
Brief Title: Paracetamol UNIFLASH for Buccal Use Phase III Trial in Acute Pain Due to a Tooth Extraction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Unither Pharmaceuticals, France (Industry)
Collaborators: AIXIAL Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UP-CLI-2020-001
Record Dates: First submitted 2020-11-16; First posted 2020-11-23 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Acute Pain
Keywords: paracetamol
MeSH Terms: conditions — Acute Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind. Participants, Investigators, and all persons involved in the conduct, data management, and analysis of the study will be fully blind to the participant's treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Paracetamol UNIFLASH 125mg (Experimental): 1 sachet Paracetamol UNIFLASH 125mg + 2 placebo capsule
  Interventions: Drug: Paracetamol Uniflash 125mg; Drug: Placebo
- Placebo (Placebo Comparator): 1 Placebo sachet + 2 placebo capsule
  Interventions: Drug: Placebo
- Paracetamol 500mg (Active Comparator): 1 Placebo sachet + 1 placebo capsule + 1 capsule Panadol 500mg
  Interventions: Drug: Panadol 500 MG Oral Tablet X1; Drug: Placebo
- Paracetamol 1000mg (Active Comparator): 1 Placebo sachet + 2 capsules Panadol 500mg
  Interventions: Drug: Panadol 500 MG Oral Tablet X2; Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol Uniflash 125mg — Oromucosal solution 1.25 mL for buccal use
  Arms: Paracetamol UNIFLASH 125mg
Drug: Panadol 500 MG Oral Tablet X1 — Tablet masked in capsule
  Arms: Paracetamol 500mg
Drug: Panadol 500 MG Oral Tablet X2 — Tablet masked in capsule
  Arms: Paracetamol 1000mg
Drug: Placebo — Dummy treatment

SUMMARY:
This study aims to evaluate the analgesic efficacy of single dose of a new paracetamol formulation (paracetamol UNIFLASH) for buccal use in comparison to two different doses of an oral paracetamol form controlled versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged from 18 years of age
* Patients scheduled to undergo the removal of one third soft-tissue impacted or not-impacted mandibular molar (associated or not to an ipsilateral erupted maxillary molar) under short-acting local anaesthetic preoperatively;
* Patients weighing > 50 kg;

Additional inclusion criteria

* Patients experiencing a moderate pain within 4 hours after the dental extraction, defined by a baseline pain intensity Visual Analogic Scale (VAS) score ≥ 40 mm and ≤ 60 mm;
* Third mandibular molar extraction completed without any immediate complication, that in the opinion of the investigator, would interfere with the study conduct and/or assessments (e.g., suspected neurosensory complication, incomplete removal of tooth).

Exclusion Criteria:

* Patient who undergoes an extraction of contralateral molar in the same procedure or a bony-impacted molar;
* Patients treated by analgesics or nonsteroidal anti-inflammatory drugs (NSAIDs) within the 3 days prior to the day of randomization (or within 5 times the elimination half-life whichever the longest);
* Patient who received other analgesic than short-acting preoperative or intraoperative local anaesthetic agents within 12 hours before the start of the surgery or peri-operatively until randomization;
* Patients with any known hypersensitivity to paracetamol, ibuprofen or ingredients contained in IMPs and Non-Investigational Medicinal Product (NIMP);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Ranked Efficacy Endpoints: 1. Sum of Pain Intensity Difference (SPID0-60min) | At 60 minutes
  Pain Intensity Difference will be calculated using the scores of pain intensity assessed by the patient at defined time-points (T5, T10, T15, T20, T30, T45, T60 min) after the IMP intake and/or right before first intake of rescue medication using a 100-mm Visual Analogic Scale (0= no pain and 100= worst imaginable pain) compared to baseline
Onset of pain relief (versus 500 mg of the reference oral paracetamol (Panadol®) | At 60 minutes
  Defined as the period for the patient to reach a meaningful pain relief during the first 60 min post-IMP intake.
  After completion of the 5-point verbal rating scale (VRS) at T5, T10, T15, T20, T30, T45, T60 min post-IMP intake assessment time points, the patient will have to answer this question "Do you consider this level of pain relief as meaningful - Yes or No?"
Proportion of responder patients at 60 minutes (versus 500 mg of the reference oral paracetamol (Panadol®)). | At 60 minutes
  A responder patient is defined as a subject who achieves a reduction of 50 % of pain intensity compared to baseline.
Patient Global Impression of Change (PGIC) versus 1000 mg of the reference oral paracetamol (Panadol®) | At 60 minutes
Onset of pain relief (versus 1000 mg of the reference oral paracetamol (Panadol®)). | At 60 minutes
  Defined as the period for the patient to reach a meaningful pain relief during the first 60 min post-IMP intake.
  After completion of the a 5-point verbal rating scale at T5, T10, T15, T20, T30, T45, T60 min post-IMP intake assessment time points, the patient will have to answer this question "Do you consider this level of pain relief as meaningful - Yes or No?"

SECONDARY OUTCOMES:
Sum of Pain Intensity Difference at 5 minutes (SPID0-5min), 10 minutes (SPID0-10min), 30 minutes (SPID0-30min), 45 minutes (SPID0-45min), 1 hour (SPID0-1h), 2 hours (SPID0-2h), 4 hours (SPID0-4h), and 6 hours (SPID0-6h). | At 5 minutes, 10 minutes, 30 minutes, 45 minutes, 1 hour, 2 hours, 4 hours, and 6 hours.
  Pain Intensity Difference will be calculated using the score of pain intensity assessed by the patient at defined time-points (T5, T10, T15, T20, T30, T45, T90, T120, T180, T240, T300 and T360 min) after IMP intake or right before first intake of rescue medication using a 100-mm Visual Analogic Scale compared to baseline.
Proportion of responders at 60 minutes (versus 1000 mg of the reference oral paracetamol (Panadol®)). | At 60 minutes
  A responder patient is defined as a subject who achieves a reduction of 50 % of pain intensity compared to baseline.
Proportion of responders at 5 minutes, 10 minutes, 30 minutes, 45 minutes, 2 hours, 4 hours and then 6 hours. | At 5 minutes, 10 minutes, 30 minutes, 45 minutes, 2 hours, 4 hours and then 6 hours.
  A responder patient is defined as a subject who achieves a reduction of 50 % of pain intensity compared to baseline at each time point of the study.
Total Pain Relief at 1 hour (TOTPAR0-1h), 2 hours (TOTPAR0-2h), 4 hours (TOTPAR0-4h) and 6 hours (TOTPAR0-6h) | At 1 hour, 2 hours, 4 hours and 6 hours.
  Pain relief (PAR) will be assessed by the patient at defined time points (T5, T10, T15, T20, T30, T45, T60, T90, T120, T180, T240, T300 and T360 min) after IMP intake and/or right before first intake of rescue medication using a 5-point verbal rating scale.
Period of time before taking rescue analgesic treatment intake. | Up to 24 hours after dose
Proportion of patients taking a rescue analgesic treatment. | At 6 hours
Patient Global Impression of Change (PGIC) versus 500 mg of the reference oral paracetamol (Panadol®) | At 60 minutes
Patient Global Impression of Change (PGIC) versus 500 mg and 1000 mg of the reference oral paracetamol (Panadol®) | At 360 minutes

OTHER OUTCOMES:
Occurrence and severity of serious and non-serious Adverse Events (AEs). | Up to 24 hours after dose
The test volume formulation acceptability | At 6 hours
  Patients will answer a question enquiring about the satisfaction with the new oromucosal solution in terms of solution volume

CONTACTS AND LOCATIONS:
Locations (20):
- France (5):
  - CHU de Bordeaux, Bordeaux
  - CHRU de Clermont Ferrand, Clermont-Ferrand
  - Hôpital Louis Mourier, Colombes
  - CHU Montpellier, Montpellier
  - CHU de Strasbourg, Strasbourg
- Italy (2):
  - Università degli Studi di Milano, Milan
  - Department of maxilla facial Surgery -University of Udine, Udine
- Poland (6):
  - University Central Stomatology GDANSK, Gdansk
  - Oral Surgery Department, Central Clinical Hospital, Lodz
  - Dental Practice, Lodz
  - Oral surgery Medical University of Lublin, Lublin
  - AW Clinic, Warsaw
  - NZOZ Akademicka Poliklinika Stomatologiczna, Wroclaw
- Spain (7):
  - Centro Médico Teknon - Grupo Quironsalud, Barcelona
  - Hospital Odontológico Universitat Barcelona, Barcelona
  - Facultad de Odontología de la Universidad de Granada, Granada
  - Instituto Profesor Sada, Madrid
  - Faculty of Medicine of the UNIVERSITY OF MURCIA, Murcia
  - Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No
At this stage, IPD sharing plan has to been discussed and finalised